CLINICAL TRIAL: NCT05853016
Title: A Urine Sample Collection Study in Apparently Healthy Adults and Adults With Chronic, Stable Morbidities
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Astute Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AST-017
Record Dates: First submitted 2023-03-09; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-03

CONDITIONS: Healthy; Chronic Disease
MeSH Terms: conditions — Chronic Disease | interventions — Urine Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (2):
- Cohort A: Healthy adults
  Interventions: Diagnostic Test: Urine collection for NEPHROCLEAR CCL14 Test
- Cohort B: Adults with stable chronic morbidities
  Interventions: Diagnostic Test: Urine collection for NEPHROCLEAR CCL14 Test

INTERVENTIONS:
Diagnostic Test: Urine collection for NEPHROCLEAR CCL14 Test — Urine will be collected and banked for future analysis with the NEPHROCLEAR CCL14 Test

SUMMARY:
The objective of this study is collect urine samples from healthy adult subjects and subjects with stable chronic morbidities for future testing to serve as controls and establish reference ranges in the development of new invitro diagnostic devices.

ELIGIBILITY:
Cohort A

Inclusion Criteria:

1. Apparently healthy adults (age > 21 years);
2. Provide written informed consent for study participation.

Exclusion Criteria:

1. Any known or suspected acute illness or condition - including acute infections - at the time of enrollment or within the previous 30 days;
2. Any known or suspected significant new onset or chronic morbid medical condition such as those listed in the inclusion criteria for Cohort B;
3. Trauma-related surgery within the last 6 months;
4. Any surgery, hospitalization or institutionalization (such as in a nursing home) during the previous 3 months;
5. Received any blood product transfusion within the previous 2 months;
6. Pregnant women or children;
7. Prisoners or institutionalized individuals;
8. Already provided a urine sample for this study.

Cohort B

Inclusion Criteria:

1. Adults (age > 21 years);
2. One or more of the following chronic, stable morbid conditions:

i. Active cancer ii. Arrhythmia (atrial fibrillation, heart block, ventricular tachycardia) iii. Chronic coagulation abnormality iv. Chronic obstructive pulmonary disease (including emphysema, chronic bronchitis, and asthma) v. Chronic pancreatitis vi. Chronic renal insufficiency vii. Congestive heart failure viii. Coronary artery disease ix. Diabetes mellitus (Type 1 or Type 2) x. Gout xi. Hyper- or hypothyroidism xii. Hyperlipidemia (includes hypercholesterolemia) xiii. Hypertension xiv. Immunocompromised xv. Inflammatory bowel disease (including Crohn's disease and ulcerative colitis) xvi. Liver cirrhosis xvii. Neuromuscular disease xviii. Peripheral vascular disease (a.k.a. peripheral artery disease) xix. Polycystic kidney disease xx. Rheumatoid arthritis xxi. Systemic Lupus Erythematosus c. Provide written informed consent for study participation.

Exclusion Criteria:

1. Any known or suspected acute illness or condition - including acute infections - at the time of enrollment or within the previous 30 days;
2. Any new onset or unstable morbidities;
3. Trauma-related surgery within the last 6 months;
4. Any surgery, hospitalization or institutionalization (such as in a nursing home) during the previous 3 months;
5. Received any blood product transfusion within the previous 2 months;
6. Pregnant women or children;
7. Prisoners or institutionalized individuals;
8. Already provided a urine sample for this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Apparently Healthy Adults and Adults With Chronic, Stable Morbidities
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Reference interval as defined by Clinical and Laboratory Standards Institute guideline EP28 for urinary C-C motif chemokine 14 concentration measured with the NEPHROCLEAR CCL14 Test within each cohort | Determined for urine sample collected at baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Cyn3rgy Research, Gresham, Oregon, United States

IPD SHARING:
Plan to Share IPD: No